CLINICAL TRIAL: NCT06179888
Title: Randomized Phase 2 Study of Iberdomide Maintenance Therapy Following Idecabtagene Vicleucel CAR-T in Multiple Myeloma Patients
Brief Title: Iberdomide Versus Observation Off Therapy After Idecabtagene Vicleucel CAR-T for Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-10541; NCI-2023-10541 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A062102 (Other: Alliance for Clinical Trials in Oncology); A062102 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2023-12-21; First posted 2023-12-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Specimen Handling; Biopsy; iberdomide; Magnetic Resonance Spectroscopy; Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (monitoring) (Active Comparator): Patients undergo disease monitoring at monthly clinic visits until disease progression. Patients also undergo bone marrow aspiration and biopsy throughout the trial, undergo collection of blood samples at screening and on study, and undergo PET/CT and/or skeletal survey x-ray, CT, or MRI at screening and then as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Patient Monitoring; Procedure: Positron Emission Tomography; Procedure: Skeletal Survey X-Ray
- Group II (iberdomide) (Experimental): Patients receive iberdomide PO QD on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy throughout the trial, undergo collection of blood samples at screening and on study, and undergo PET/CT and/or skeletal survey x-ray, CT, or MRI at screening and then as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Iberdomide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Skeletal Survey X-Ray

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo PET/CT and/or CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Iberdomide — Given PO
  Other Names: CC 220; CC-220
  Arms: Group II (iberdomide)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Patient Monitoring — Undergo disease monitoring
  Other Names: medical monitoring; monitor
  Arms: Group 1 (monitoring)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Skeletal Survey X-Ray — Undergo skeletal survey x-ray
  Other Names: Skeletal Survey

SUMMARY:
This phase II trial compares iberdomide maintenance therapy to disease monitoring for improving survival in patients who have received idecabtagene vicleucel (a type of chimeric antigen receptor T-cell [CAR-T] therapy) for multiple myeloma. The usual approach after treatment with idecabtagene vicleucel is to monitor the multiple myeloma without giving myeloma medications. There is currently no medication approved specifically for use after idecabtagene vicleucel treatment. Upon administration, iberdomide modifies the immune system and activates immune cells called T-cells, which could enhance the effectiveness of idecabtagene vicleucel. Iberdomide may keep multiple myeloma under control for longer than the usual approach (disease monitoring) after idecabtagene vicleucel, and may help multiple myeloma patients live longer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish and confirm the safety and dose of iberdomide as maintenance after idecabtagene vicleucel (ide-cel) CAR-T. (Safety run-in) II. To assess whether iberdomide maintenance therapy after idecabtagene vicleucel CAR-T cell therapy increases progression-free survival (PFS) relative to observation without additional therapy. (Randomized phase II)

SECONDARY OBJECTIVES:

I. To demonstrate anti-tumor activity, defined as conversion from non-minimal residual disease (MRD) complete response (CR)/stringent CR (sCR) status to MRD-negative CR/sCR, as well as improvement in PFS in the safety run-in cohort. (Safety run-in) II. To estimate the rate of conversion from MRD-positive at baseline to MRD-negative at any time point post-initiation of iberdomide maintenance or observation without additional therapy. (Key secondary objective; Randomized phase II) III. To estimate overall survival (OS) distribution post-initiation of iberdomide maintenance or observation without additional therapy. (Key secondary objective; Randomized phase II) IV. To estimate the minimal residual disease (MRD)-negativity rate at pre-registration and at one year post-initiation of iberdomide maintenance or observation without additional therapy. (Randomized phase II) V. To estimate rate of deepening hematological response among patients with measurable multiple myeloma (MM) post-initiation of iberdomide maintenance or observation without additional therapy. (Randomized phase II) VI. To evaluate the safety profile of iberdomide maintenance. (Randomized phase II) VII. To evaluate the peripheral blood immunophenotype before and during iberdomide maintenance or observation without additional therapy. (Randomized phase II) VIII. To evaluate persistence of CAR-T cells with iberdomide maintenance or observation without additional therapy. (Randomized phase II)

CORRELATIVE SCIENCE OBJECTIVES:

I. To estimate the minimal residual disease (MRD)-negativity rate at start of maintenance and at one year post-initiation of maintenance or observation.

II. To estimate the sustained MRD-negativity rate. III. To estimate the rate of conversion from MRD-positive to MRD-negative. (Key objective) IV. To evaluate the peripheral blood immunophenotype before and during maintenance therapy or observation.

V. To evaluate the persistence of CAR-T cells. VI. To evaluate B-cell maturation antigen (BCMA) protein expression by immunohistochemistry on myeloma cells from patients that have relapsed/recurrent disease.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP 1: Patients undergo disease monitoring at monthly clinic visits until disease progression. Patients also undergo bone marrow aspiration and biopsy throughout the trial, undergo collection of blood samples at screening and on study, and undergo positron emission tomography (PET)/computed tomography (CT) and/or skeletal survey x-ray, CT, or magnetic resonance imaging (MRI) at screening and then as clinically indicated.

GROUP 2: Patients receive iberdomide orally (PO) once daily (QD) on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy throughout the trial, undergo collection of blood samples at screening and on study, and undergo PET/CT and/or skeletal survey x-ray, CT, or MRI at screening and then as clinically indicated.

After completion of study treatment, patients are followed up within 30 days, then every 3-6 months until 4 years following registration.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION ELIGIBILITY CRITERIA (STEP 0):
* All patients must be pre-registered. For patients who consent to biobanking, submit the bone marrow and blood specimens

  * Note: Patients who do not consent to the optional biobanking must be pre-registered, but specimens should not be submitted for these patients
  * Please ensure patient has suspected diagnosis of multiple myeloma and meets on study guidelines prior to informed consent and biospecimen collection
  * In cases where the bone marrow aspiration may be inadequate at Step 0 registration, the patient may still register on study
* ELIGIBILITY CRITERIA (STEP 1):
* Patients must have diagnostically confirmed MM in response status of stable disease or better by International Myeloma Working Group (IMWG) criteria at day 80-110 post-infusion of ide-cel. Patients in deep remission (e.g., CR, MRD-negative, etc.), are eligible
* All patients are required to have received ide-cel CAR-T within 80-110 days of registration
* Adverse events related to ide-cel are required to have resolved to grade =< 1 except fatigue, alopecia, and other events that are unlikely to interfere with study assessments or pose a safety risk to participants
* Patients must have had ≥ 4 lines of therapy for MM (this includes proteasome inhibitor, immunomodulatory agent, and anti-CD38 monoclonal antibody)
* Prior therapy with iberdomide is permitted but prior iberdomide refractoriness is prohibited. Refractoriness is defined as per published IMWG criteria; progression while on iberdomide or within 60 days of stopping iberdomide
* Patients who have received MM-directed therapy since ide-cel infusion are not eligible, with the exception of short-course steroids for managing ide-cel toxicity as described below
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3

  * Platelet transfusions or use of growth factors for neutropenia (e.g., filgrastim, tbo-filgrastim, sagramostim) are not permitted to meet enrollment criteria
* Platelet count ≥ 75,000/mm^3

  * Platelet transfusions or use of growth factors for neutropenia (e.g., filgrastim, tbo-filgrastim, sagramostim) are not permitted to meet enrollment criteria
* Calculated (calc.) creatinine clearance >= 30 mL/min by Modification of Diet in Renal Disease (MDRD)

  * Platelet transfusions or use of growth factors for neutropenia (e.g., filgrastim, tbo-filgrastim, sagramostim) are not permitted to meet enrollment criteria
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)

  * Platelet transfusions or use of growth factors for neutropenia (e.g., filgrastim, tbo-filgrastim, sagramostim) are not permitted to meet enrollment criteria
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 3 x upper limit of normal (ULN)

  * Platelet transfusions or use of growth factors for neutropenia (e.g., filgrastim, tbo-filgrastim, sagramostim) are not permitted to meet enrollment criteria
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effect on the developing fetus and newborn are unknown.

  * FCBP (female of childbearing potential) is a female who: 1) has achieved menarche (first menstrual cycle) at some point, 2) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time during the preceding 24 consecutive months).
  * Females of childbearing potential (FCBP):

    * Must use a contraceptive method that is highly effective (with a failure rate of < 1% per year), preferably with low user dependency during the intervention period and for at least 28 days after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.
    * The effects of iberdomide on the developing human fetus are unknown. Immunodulatory derivative (IMiD) agents as well as other therapeutic agents used in this trial are known to be teratogenic. Females of child-bearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to, and again within 24 hours of starting iberdomide, and must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control, one highly effective method and one additional effective method at the same time, at least 28 days before she starts taking iberdomide. Examples of highly effective methods are intrauterine device, hormonal contraceptives, tubal ligation, or partner's vasectomy. Examples of barrier method are male condom, diaphragm, or cervical cap. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risk of fetal exposure.
    * Should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study, she should inform her treating physician immediately. FCBP must use adequate contraception for at least 28 days after discontinuation from study. Because of the potential for serious adverse reactions in a breastfed child, women are advised not to breastfeed during treatment and for at least 28 days after the last dose.
    * The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with a nearly undetected pregnancy.
  * Non-childbearing potential is defined as follows (by other than medical reasons):

    * ≥ 45 years of age and has not had menses for > 1 year
    * Patients who have been amenorrhoeic for < 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
    * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure
* Male patients must agree to use an adequate method of contraception for the duration of the study and for 28 days afterwards.

  * Male participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies:

    * Male participants are eligible to participate if they agree to the following during the intervention period and for 28 days after the last dose of study treatment to allow for clearance of any altered sperm:

      * Refrain from donating sperm

PLUS, either:

* Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
* Must agree to use contraception/barrier as detailed below:

  * Agree to use a male condom, even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of < 1% per year as when having sexual intercourse with a woman of childbearing potential (including pregnant females)

    * Patients may not have polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome or amyloidosis involving any vital organ; amyloidosis found in skin or lymph nodes ("non-vital organs"), or incidental observation of amyloidosis on bone marrow biopsy, are both permissible. Plasma cell leukemia is permissible for study enrollment
    * Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
    * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration are eligible for this trial
    * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
    * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. Patients with HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load
    * Patients may not have other, active infections at time of study registration. Recent infections are not exclusionary if antibiotics have been completed and infection is considered to be resolved / controlled. (Chronic maintenance antibiotics for prior infections, such as fungal, are permissible.)
    * No known allergy to iberdomide
    * No known medical condition causing an inability to swallow oral formulations of agents
    * Patients receiving other active therapies for MM since ide-cel infusion are prohibited from participating in the study
    * Corticosteroids used for the purpose of managing ide-cel toxicity (often neurotoxicity) soon after ide-cel administration are acceptable, provided that the participant will have been off corticosteroids for > 30 days by cycle 1 day 1. Physiologically dosed chronic steroids are permitted
    * Given the potential for interaction with iberdomide, patients who take strong CYP3A4 inducers or inhibitors may enroll after switching to a different agent and after an appropriate washout period for that particular medication, ideally three half-lives, prior to cycle 1 day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (safety run-in) | The first 3 months of therapy
Progression-free survival (PFS) (randomized phase II) | From randomization to the time of progression and/or death, assessed up to 4 years
  Final analyses will use log-rank test statistics to compare the PFS distributions between the treatment arms. Will also evaluate differences in PFS between the treatment arms using a stratified log-rank test. In addition, the methods of Kaplan and Meier will be used to graphically evaluate these distributions as well as to estimate the median PFS and corresponding 95% confidence intervals. Further, will also estimate the 1- and 2-year PFS rates for each treatment arm along with corresponding 95% confidence intervals. Finally, Cox proportional hazards models will be used to evaluate the impact of treatment arm on PFS.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 4 years
  Adverse events will be collected and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 criteria. For CTCAE data, the maximum grade for each type of adverse will be recorded for each patient, and described using frequency tables. All-cause adverse events will be summarized as well as treatment-related adverse events, with particular focus on grade 3+ non-hematologic adverse events and grade 4+ hematologic events. Frequency tables will be reviewed to identify patterns. The overall adverse event severity will be compared between treatment arms using a chi-square test (or Fisher's exact test if the data in contingency table is sparse).
Number of treatment cycles received (tolerability) | Up to 4 years
  Will be summarized.
Proportion of patients with dose modifications, omissions, and/or delays (tolerability) | Up to 4 years
  Will be summarized.
Proportion of patients who go off treatment due to adverse events | Up to 4 years
  Will be summarized.
Overall survival (OS) | From randomization until death from any cause, assessed up to 4 years
  The Kaplan-Meier method will be used to estimate OS for each treatment arm, with 1- and 2-year OS estimates and OS medians along with their 95% confidence intervals. For the comparison of the treatment arms, will use a one-sided log-rank test to compare the OS distributions between treatment arms. Will also evaluate the influence of arm on OS using stratified and unstratified multivariable Cox proportional hazards models.
Best response achieved while on study | Up to 4 years
  Will calculate these rates by treatment arm along with corresponding 95% binomial confidence intervals. Logistic regression models may also be used to assess differences in the ability to deepen or convert to a response between treatment arms. Minimal residual disease (MRD) will be assessed as an aspect of response assessment.
Proportion of patients who improve their status | After randomization, up to 4 years
  Will calculate these rates by treatment arm along with corresponding 95% binomial confidence intervals. Logistic regression models may also be used to assess differences in the ability to deepen or convert to a response between treatment arms. MRD will be assessed as an aspect of response assessment.

OTHER OUTCOMES:
MRD-negativity rate | At start of maintenance and at one year post-initiation of maintenance or observation
  Will evaluate and identify patients in MRD-negative complete response (CR)/stringent CR (sCR) versus patients who are not in MRD-negative CR/sCR, both from pre-registration (before start of maintenance iberdomide vs. active monitoring) and at the follow-up time points. These will be summarized as proportions within each of the randomization arms at each time point. Assuming that the number of MRD-negative CR/sCR patients is binomially distributed, will calculate corresponding 95% binomial confidence intervals for these rates as well.
Sustained MRD-negativity rate | Up to 4 years
  Will evaluate and identify patients in MRD-negative CR/sCR versus patients who are not in MRD-negative CR/sCR, both from pre-registration (before start of maintenance iberdomide vs. active monitoring) and at the follow-up time points. These will be summarized as proportions within each of the randomization arms at each time point. Assuming that the number of MRD-negative CR/sCR patients is binomially distributed, will calculate corresponding 95% binomial confidence intervals for these rates as well.
Rate of conversion from MRD-positive to MRD-negative | Up to 4 years
  Will assess the proportion of patients who had detectable disease at randomization who were able to achieve MRD-negative CR/sCR status after treatment with iberdomide.
Peripheral blood immunophenotype | Before and during maintenance therapy or observation
  Continuous measures of immune cell subsets will be evaluated using side-by-side boxplots to show differences between treatment arms, and two-sample t-tests will be used to assess quantitative differences in the mean levels of these measures between arms.
Persistence of chimeric antigen receptor T-cells | At cycle 12
B-cell maturation antigen (BCMA) protein expression | Up to 4 years
  Will evaluate protein expression by immunohistochemistry on myeloma cells from patients that have relapsed/recurrent disease. Will summarize the BCMA expression status at baseline and evaluate how these associate with PFS using Cox regression models, to evaluate how treatment arm may modify this influence. Changes in this status can be captured both graphically as well as a time-dependent covariate in the model for PFS. In a similar manner, will also evaluate expression intensity. This will be done in those with BCMA expression present, but also across all patients. Differences in changes in these expression intensity levels before versus after study registration monitoring will be compared between treatment arms. Changes in this status will also be evaluated and how these may differ between patients treated with maintenance iberdomide vs. active monitoring using logistic generalized estimating equation models.

CONTACTS AND LOCATIONS:
Overall Officials: Sascha A Tuchman, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (73):
- United States (73):
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Augusta University Medical Center, Augusta, Georgia
  - University of Illinois, Chicago, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Levine Cancer Institute - Huntersville, Huntersville, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Houston Methodist San Jacinto Hospital, Baytown, Texas
  - Houston Methodist Cypress Hospital, Cypress, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm